CLINICAL TRIAL: NCT04602962
Title: Studies Aiming at Identifying Predictors for Fertility Treatments' Outcomes and to Evaluate the Efficacy and Safety of Fertility Preservation
Brief Title: Efficacy and Safety of Fertility Treatments and Fertility Preservation
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Kenny Rodriguez-Wallberg, MD, PhD, Associate Professor, Karolinska Institutet
Other Study IDs: KI-KRW-200909-201505
Record Dates: First submitted 2015-05-18; First posted 2020-10-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Infertility
Keywords: fertility preservation; fertility treatment; safety; efficacy; fertility outcomes; follow-up; cohort
MeSH Terms: conditions — Infertility | interventions — Fertility Preservation; Cryopreservation; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fertility preservation performed: subgroup analysis by cause of infertility, clinical characteristics, biochemical markers
  Interventions: Procedure: fertility preservation, several methods
- Fertility preservation not performed: subgroup analysis by cause of infertility, clinical characteristics, biochemical markers

INTERVENTIONS:
Procedure: fertility preservation, several methods — fertility preservation using assisted reproductive techniques or not
  Other Names: cryopreservation, surgery
  Groups: Fertility preservation performed

SUMMARY:
This study analyses clinical data prospectively collected for over a decade in several clinical databases. Electronic medical records are available since 1998.

Since 2011 the subgroup of patients that undergo fertility preservation are invited to participate in a prospective study aiming at long-term follow-up after fertility preservation for oncologic and non-oncologic conditions.

DETAILED DESCRIPTION:
In this study, the investigators aim at analyze the treatment outcomes of patients with infertility, their clinical characteristics and biochemical parameters aiming at identifying predictors for the treatment outcomes.

For the cohort of patients that have undergone fertility preservation at Karolinska University Hospital, the investigators aim at investigating efficacy and safety of the procedures.

The data can be expanded by using additional databases such as the Regional Cancer Registry and other registries.

Analysis of data collected will allow the investigation of efficacy and safety of fertility preservation, identification of predictors for fertility outcomes,prediction of future activities and costs of the procedures.

ELIGIBILITY:
Inclusion Criteria:

* infertile patients and patients who undergo fertility preservation

Exclusion Criteria:

* Healthy individuals, fertile population

Max Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cohort collected from the registers of the university hospitals of Sweden, each representing a health care region, from 1995 and ongoing. FP is included in the tax funded healthcare system and data is registered all over the country. Date is also compared with the Swedish tax registry.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2009-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy and safety of fertility preservation - Long-term follow-up | 2028
  Correlation between method of fertility preservation and pregnacy rate

SECONDARY OUTCOMES:
Clinical outcome of fertility treatments i breast cancer patients | 5-20 years post diagnosis
  Fertility treatment vs no fertility treatment i breastcancer patients: effect on survival
Clinical outcome of fertility treatments i breast cancer patients | 5-7 years post diagnosis
  Fertility treatment vs no fertility treatment i breastcancer patients: effect on disease free survival
Predictors of effictive fertility treatment | patient data collected from time of treatment, pregnancy rate until end of study
  Correlation between clinical variables (age, BMI, oocyte level, administered gonadotropins, infertility) method of fertility preservation and Pregnancy rate
Efficacy and safety of COS using GnRHa for fertility preservation in BC patients | Observed outcomes in patients registered between 1995 and 2017. Follow up until end of 2018.
  hCG vs GnRH trigger on effect on number of cryopreserved embryos and oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Dan Grandér, Prof, Study Chair — Karolinska Institutet
Locations (1):
- Reproductive Medicine, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wikander I, Lundberg FE, Nilsson H, Borgstrom B, Rodriguez-Wallberg KA. A Prospective Study on Fertility Preservation in Prepubertal and Adolescent Girls Undergoing Hematological Stem Cell Transplantation. Front Oncol. 2021 Jun 30;11:692834. doi: 10.3389/fonc.2021.692834. eCollection 2021. PMID 34277437